CLINICAL TRIAL: NCT06692179
Title: An Open-Label, Pilot Clinical Trial To Test The Safety And Feasibility Of A Suspension of Freeze-dried Microbiota In Patients Undergoing Colon Resection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Freeze-dried Microbiota
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Clostridioides Difficile Infection; Colonic Surgery
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Intervention Model Description: This Phase 1 pilot clinical trial that will evaluate the initial safety and feasibility of orally administered preparation of fecal microbiota (MTP-101P) in patients undergoing colon resection.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Male and female patients, ages 18-75, diagnosed with colon polyps or early (stage I or II) colorectal cancer or medically refractory diverticulitis.
  Interventions: Drug: Orally administered preparation of fecal microbiota (MTP-101P)

INTERVENTIONS:
Drug: Orally administered preparation of fecal microbiota (MTP-101P) — As per standard of care, patients will receive MBP and OA the day prior to surgery as well as IV antibiotics at the time of surgery. MTP-101P will be given 48 hours after the administration of the dose of IV antibiotics to avoid the undesired bactericidal effects of antibiotics on the bacterial load from MTP-101P.

SUMMARY:
This Phase 1 pilot clinical trial that will evaluate the initial safety and feasibility of orally administered preparation of fecal microbiota (MTP-101P) in patients undergoing colon resection. We plan to enroll male and female patients, ages 18-75, diagnosed with colon polyps or early (stage I or II) colorectal cancer or medically refractory diverticulitis. We will recruit 40 patients total to receive the investigational product. This trial will inform development of future trials in treatment of colon and rectal surgery. Active drug is composed of highly purified, freeze-dried, fecal microbiota from healthy donors. This study will also allow for limited evaluation of pharmacokinetics in terms of donor microbiota engraftment. The exploratory objective is to evaluate engraftment of donor microbiota with this preparation and compare the results with data generated with the data generally from microbiota transplantation (IND28152). Stool samples may be returned via mail rather than clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Able/willing to provide informed consent
* Between 18-75 years of age
* Undergoing surgery for unresectable polyps, early-stage colon cancer (Stage 1 or 2) not predicted based on pre-operative National Comprehensive Cancer Network guidelines to meet criteria for adjuvant chemotherapy, or a history of diverticulitis.
* Able to provide fecal samples.
* Stated willingness to comply with all study procedures and availability for the duration of trial to follow-up by telephone, in-person, email, and/or video visits or correspondence

Exclusion Criteria:

* Any history of inflammatory bowel disease
* Pregnancy or breastfeeding. A pregnancy test will be obtained from females of child-bearing potential on the proposed day of MTP-101P (prior to its administration). Patients with a positive pregnancy test will be excluded. A negative result will be required for subjects who are females of child-bearing potential to receive MTP-101P.
* Life expectancy of < 6 months
* Presence of ileostomy or colostomy
* Known history of inflammatory bowel disease (Crohn's, Ulcerative Colitis)
* Patients on immunosuppressants (calcineurin inhibitors, prednisone ≥ 20 mg/day, methotrexate, azathioprine, immunosuppressive biologics, JAK inhibitors).
* Patients with neutropenia (an absolute neutrophil count <0.5 x 10^9 cells/L) obtained on a complete blood count with differential at screening.
* History of solid organ or bone marrow transplant.
* Anticipated recurrent antibiotic use (e.g., patients with frequent urinary tract infections or sinusitis).
* History of severe anaphylactic food allergy.
* History of celiac disease.
* Patients receiving cancer chemotherapy, immunotherapy, or radiation.
* Subjects who, in the opinion of the Investigator, are not capable of giving informed consent for the study or who are unable or unwilling to adhere to the study requirements outlined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-02-18 (Estimated); Study Completion 2027-02-18 (Estimated)

PRIMARY OUTCOMES:
Evaluate engraftment of donor microbiota (see 15.3 for statistics) via determination of alpha and beta diversity. | Day180
  (via alpha and beta diversity statistics) essentially compares the study patient's microbiome composition at any time point when stool is collected to the microbiome composition of the donor fecal transplant that the study patient receives. Before receiving the fecal transplant, we do not expect the study patient's microbiome composition to mirror the donor. However, after giving the donor fecal transplant, we expect the study patient's microbiome composition to look similar to the transplant they were given.
Compare baseline microbiome characteristics with changes over time after MTP-101P. | Day180
  In addition to the microbiome compositional statistics we will calculate that are detailed above, we will assess measures of gut health and immune function before and after receiving the fecal transplant. These will be the quantity of short-chain fatty acids in the stool, gut barrier markers in the serum (CD-14, occludin, ZO-1), and overall immune function.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus Jahansouz, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States